CLINICAL TRIAL: NCT01620710
Title: Hypofractionated Helical Intensity-Modulated Radiotherapy of the Prostate Bed After Prostatectomy With or Without the Pelvic Lymph Nodes - the PRIAMOS Trial
Brief Title: Safety Study of a Shorter (Hypofractionated) Radiotherapy for the Prostate Bed With or Without the Pelvic Lymph Nodes
Acronym: PRIAMOS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Klaus Herfarth, MD, Principal Inverstigator, Heidelberg University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRIAMOS
Record Dates: First submitted 2012-06-13; First posted 2012-06-15 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Prostate Cancer
Keywords: prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- prostate bed (Other): irradiation of the prostatic bed only (no higher risk of lymph node recurrence); helical IMRT of the prostate bed (18 x 3 Gy)
  This arm has already finished recruitment
  Interventions: Radiation: hypofractionated helical IMRT
- prostate bed & lymph nodes (Other): irradiation of the prostatic bed and the pelvic lymphatic drainage (in patients with higher risk of lymph node recurrence); helical IMRT of the prostate bed (18 x 3 Gy) and the pelvic lymph nodes (18 x 2.5 Gy)
  Interventions: Radiation: hypofractionated helical IMRT

INTERVENTIONS:
Radiation: hypofractionated helical IMRT — hypofractionated helical IMRT of the prostate bed, 18 x 3 Gy
Radiation: hypofractionated helical IMRT — helical IMRT of the prostate bed (18 x 3 Gy) and the pelvic lymph nodes (18 x 2.5 Gy)

SUMMARY:
This trial investigates safety and feasibility of a hypofractionated radiotherapy (i.e. with higher daily doses and shorter total treatment time compared to standard fractionation) of the prostate bed with or without the pelvic lymph nodes.

DETAILED DESCRIPTION:
While evidence on safety and efficacy of primary hypofractionated radiotherapy in prostate cancer is accumulating, data on postoperative hypofractionated treatment of the prostate bed and of the pelvic lymph nodes is still scarce. This phase II trial was initiated to investigate safety and feasibility of hypofractionated treatment of the prostate bed alone or with the pelvic lymph nodes.

A total of 80 prostate cancer patients with the indication for adjuvant radiotherapy will be enrolled, where 40 patients with a low risk of lymph node involvement (arm 1) and another 40 patients with a high risk of lymph node involvement (arm 2) will each receive 54 Gy in 18 fractions to the prostate bed. Arm 2 will be given 45 Gy to the pelvic lymph nodes additionally. Helical Tomotherapy and daily image guidance wil be used.

ELIGIBILITY:
Inclusion Criteria:

* resected prostate carcinoma with histological grading (Gleason Score)
* status post prostatectomy for a pT3 carcinoma and/or R1/2 resection or PSA recurrence after prostatectomy (2 consecutive PSA rises)
* PSA recurrence ≥ 1 ng/ml: CT/PET/MRI imaging excluding pathological lymph nodes
* Karnofksy performance score ≥ 70 %
* age 18 - 80 years
* only arm 2: antihormonal therapy for 2 months prior to radiotherapy and continuation of hormonal suppression after radiotherapy recommended
* written informed consent

Exclusion Criteria:

* patient's refusal
* patient's inabillity to give informed consent
* stage IV (distant metastases)
* lymph node involvement outside the pelvis
* severe wound complications after laparatomy
* only arm 2: severe lymphoedema of the legs, elephantiasis, postthrombotic syndrome
* decompensated pulmonary, cardiovascular, metabolic, hematopoetic, coagulatory or renal comorbidities
* known other malignant disease with distant metastases
* prior pelvic irradiation
* participation in another clinical trial that might compromise the results of the PRIAMOS trial or the other trial

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
proportion SDR of patients with no grade III/IV toxicity and/or treatment discontinuation | 2 years
  Proportion SDR of patients with no NCI CTC AE grade 3-4 toxicity and no discontinuation of treatment during the full set of 18 fractions by any reasons in the intent-to-treat (ITT) population

SECONDARY OUTCOMES:
biochemical recurrence free survival (BFS) | 2 years
Quality of Life | 2 years
  Quality of Life Scores as measured by the EORTC-QLQ30 and -PR25 questionnaires
overall survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Herfarth, MD, Principal Investigator — Heidelberg University
Locations (1):
- Dep. of Radiation Oncology, University Hospital of Heidelberg, Heidelberg, Germany

REFERENCES:
- [Result] Katayama S, Striecker T, Kessel K, Sterzing F, Habl G, Edler L, Debus J, Herfarth K. Hypofractionated IMRT of the prostate bed after radical prostatectomy: acute toxicity in the PRIAMOS-1 trial. Int J Radiat Oncol Biol Phys. 2014 Nov 15;90(4):926-33. doi: 10.1016/j.ijrobp.2014.07.015. Epub 2014 Sep 9. PMID 25216858
- [Derived] Krause S, Sterzing F, Neuhof D, Edler L, Debus J, Herfarth K. Hypofractionated helical intensity-modulated radiotherapy of the prostate bed after prostatectomy with or without the pelvic lymph nodes - the PRIAMOS trial. BMC Cancer. 2012 Oct 31;12:504. doi: 10.1186/1471-2407-12-504. PMID 23114055